CLINICAL TRIAL: NCT02957760
Title: Prevention of Retinal Non-perfusion in Central Retinal Vein Occlusion by Hydroxycarbamide Treatment.
Acronym: PNPRO_HC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Hopital Universitaire Robert-Debre (Other); Institut National de la Transfusion Sanguine (Other); Keyrus Biopharma (Other); For Drug Consulting (Other); Theravia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P15-01
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Central Retinal Vein Occlusion, Non-Ischemic
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hydroxycarbamid — 20 mg/kg milligram(s)/kilogram per day during 6 month, oral administration (coated tablet).
  Other Names: siklos

SUMMARY:
The central retinal vein occlusion (CRVO) is a major cause of ocular morbidity, depending in particular on the occurrence and extent of retinal ischemia by capillary occlusion. There is no effective systemic treatment of this condition. An increase in the adhesion of erythrocytes to vascular endothelium was observed for patients with CRVO, correlated with overexpression of membrane phosphatidylserine

DETAILED DESCRIPTION:
introduction : The central retinal vein occlusion (CRVO) is a major cause of ocular morbidity, depending in particular on the occurrence and extent of retinal ischemia by capillary occlusion. There is no effective systemic treatment of this condition. An increase in the adhesion of erythrocytes to vascular endothelium was observed for patients with CRVO, correlated with overexpression of membrane phosphatidylserine.

Hypothesis : Hydroxycarbamide (HC) by reducing the erythrocyte adhesion to the endothelium may prevent or delay the onset of retinal capillary non-perfusion in patients with CRVO.

Primary objective: To assess the efficacy at 3 months of treatment with HC on retinal capillary perfusion in patients with a recent CRVO.

Secondary Objectives: To evaluate the safety of the treatment, the efficacy to 6 months on retinal perfusion of the treatment with HC (HC peak effect on the red cell adhesion in vitro), and the biological effects of HC, in particular on adhesion to endothelium and erythrocyte hemorheological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes of at least 45 years of age.
* with social protection
* Presenting CRVO for less than 1 month duration
* With a decrease of visual acuity and with the best corrected visual acuity lower than 6/10 (73 ETDRS letters)
* Signature of informed consent

Exclusion Criteria:

* predictable lack of compliance to the protocol
* monophtalmic patient or any ocular history or condition that could interfere with the study course or results interpretation.
* active systemic disease
* sickle cell disease
* myeloproliferative disease
* myelosuppression
* kidney or liver insufficiency
* ongoing treatment with hydroxycarbamide or anticoagulant
* Pregnancy, breast-feeding, no efficient contraception (for both sexes)
* wish of paternity (for males of al least 45 years of age)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
retinal capillary non-perfusion | 3 months
  To assess the percentage of subjects in whom one of the following events will not be observed at W13 (any event being considered as one of the criteria of worsening of retinal capillary non-perfusion):
  * Occurence of at least one direct sign of retinal ischemia: Increase of more than 30% of peripheral retinal non-perfusion on large-field angiography or of the central avascular zone of the retina,
  * Occurence of at least one indirect sign of retinal ischemia: reperfusion of the aterial iris circle, rubeosis iridis, neovascular glaucoma or abolition of the afferent pupillary reflex.

SECONDARY OUTCOMES:
retinal capillary non-perfusion | 2 weeks, 2 months and 6 months
  Same criteria of retinal non perfusion as for primary end point
Hydroxycarbamide safety - visual acuity and retinal thickness. Biological in vitro effects on erythrocyte adhesion to vascular endothelium and various haemorheological parameters. | 2 weks, 2 months, 3 months and 6 months
  HC effect on visual acuity and retinal thickness. Biological in vitro effects on erythrocyte adhesion to vascular endothelium and various haemorheological parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Girmens, Principal Investigator — CHNO des Quinze-Vingts
Locations (1):
- CHNO des Quinze-Vingts, Paris, France